CLINICAL TRIAL: NCT07297888
Title: Gabpentin vs Clonidine for Post Operative Pain
Brief Title: COMPARISON OF EFFECTS OF GABAPENTIN AND CLONIDINE ON POST-OPERATIVE PAIN AND ANXIETY IN LUMBAR SPINAL SURGERY.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shri Guru Ram Rai Institute of Medical and Health Sciences (Other)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, ABabu, All India Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2025-11-19; First posted 2025-12-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain
Keywords: gabapentin; clonidine; pain
MeSH Terms: conditions — Pain | interventions — Gabapentin; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- clonide (Active Comparator): In this group the investigators have given clonidine to the participants
  Interventions: Drug: Gabapentin
- placebo (Placebo Comparator): in this group no active drug was given to the participants
  Interventions: Drug: Gabapentin
- gabapentin (Active Comparator): In this group the investigators have given gabapentin to the participants
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — comparison of both these drugs to decrease pain
  Other Names: clonidine

SUMMARY:
the investigators have tested whether gabapentin is superior to clonidine top decrease the post operative pain during spinal surgeries as a part of their thesis study. the investigators are registering this study post date as the student forgot by mistake to do so.

ELIGIBILITY:
Inclusion Criteria:

- Eligible participants were aged 18-60 years, classified as ASA physical status I or II, and scheduled for one or two-level lumbar laminectomy.

Exclusion Criteria:

* Patients with psychiatric disorders, autoimmune diseases, local infection, BMI >35, emergency procedures, tumour surgeries and the patients requiring the postoperative ventilation were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
post operative pain | 1, 2, 4, 6, 8, 12, and 24 hours postoperatively.
  Pain was assessed using the Visual Analog Scale (VAS) score ranging from 0 to 10. 10 being the worst pain and 0 being No pain

SECONDARY OUTCOMES:
anxiety | 1, 2, 4, 6, 8, 12, and 24 hours postoperatively.
  anxiety was evaluated using Hamilton Anxiety Rating Scale (HAM-A). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Adabala Vijay Babu, Dehradun, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Yes
we can share our research question and methodology whenever it is necessary
Supporting Information: Study Protocol